CLINICAL TRIAL: NCT03030612
Title: A Phase I/II, Open-label, Dose-Escalating Study With a Proof of Concept Cohort to Evaluate the Safety, Tolerability and Efficacy of ARGX-110 in Combination With Azacytidine in Subjects With Newly Diagnosed Acute Myeloid Leukemia (AML) or High Risk Myelodysplatic Syndrome (MDS)
Brief Title: A Study of ARGX-110 in Combination With Azacytidine in Participants With Newly Diagnosed Acute Myeloid Leukemia (AML) or High Risk Myelodysplatic Syndrome (MDS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OncoVerity, Inc. (Industry)
Collaborators: argenx (Industry); Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108756; 2016-002151-17 (EudraCT Number); ARGX-110-1601 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- ARGX-110 with Azacytidine (AZA) (Experimental): Phase 1: Participants will receive loading dose of ARGX-110 1 milligram per kilogram (mg/kg) body weight (cohort 1), 3 mg/kg body weight (cohort 2), 10 mg/kg body weight (cohort 3) or 20 mg/kg body weight (cohort 4) administered intravenously (IV) in combination with AZA standard dose of 75 milligram per meter square (mg/m^2) body surface area (BSA) administered subcutaneously (SC) / intravenously (IV). Phase 2: Participants will receive loading dose of ARGX-110 IV at a recommended dose for Phase 2 (RP2D) level from phase 1 in combination with AZA standard dose of 75 mg/m^2 BSA, administered SC/IV as per local practice.
  Interventions: Drug: ARGX-110; Drug: AZA

INTERVENTIONS:
Drug: ARGX-110 — ARGX-110 will be administered intravenously.
  Other Names: Cusatuzumab; JNJ-74494550
Drug: AZA — AZA will be administered subcutaneously/intravenously.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of ARGX-110 and/or the recommended Phase II dose (RP2D) in combination with a standard dose of azacytidine (AZA) in Phase 1; and to evaluate efficacy of ARGX-110 when administered at a RP2D level established in Phase I in combination with a standard dose of AZA (proof-of concept) by evaluating overall response rate (ORR) in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) indicating an understanding of the purposes, risks, and procedures required for the study and willingness and ability to participate in the study
* Acute myeloid leukemia (AML) or high risk myelodysplastic syndrome (MDS) (according to 2016 World Health Organization [WHO] classification definition of greater than or equal to [>=] 20 percent [%] blasts) (bone marrow) unsuitable for intensive treatment (including stem cell transplantation) with a curative intent, but eligible to receive azacytidine (AZA) treatment
* Expected life expectancy >= 3 months, at the discretion of the investigator
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Women of childbearing potential having a negative serum pregnancy test at screening and within 48 hours before infusion of ARGX-110 on Day -14, and willing to use an effective contraceptive method (intrauterine devices, hormonal contraceptives, contraceptive pill, implants, transdermal patches, hormonal vaginal devices, infusions with prolonged release) during the study and for at least 3 months after the last study drug administration

Exclusion Criteria:

* Prior or concurrent malignancy, except for the following: (1) adequately treated basal cell or squamous cell skin cancer; (2) carcinoma in situ of the cervix; (3) carcinoma in situ of the breast; (4) incidental histological finding of Prostate cancer (Tumour, Node, Metastasis [TNM] stage T1a or T1b), or; (5) Any other cancer from which the subject has been disease-free for more than 2 years
* Any previous AML or MDS chemo- or radiotherapy (with the exception of hydroxyurea/Litalir for leukocyte control which should be discontinued by the first day of AZA, local radiation therapy, therapy for basal or squamous cell carcinoma of the skin)
* Treatment with any investigational product within 4 weeks before the first administration of ARGX-110
* Any known active or chronic infection, including human immunodeficiency virus (HIV) and hepatitis B or C virus infection
* Any other concurrent disease or medical condition that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Phase 1: Number of Participants with Dose Limiting Toxicity (DLT) | Up to 3.6 years
  DLTs will be defined as any of the following drug-related events: Any grade 3 or higher drug related non-hematological toxicity or; Grade 3 or higher IRRs or; inability to administer the next dose due to a drug-related adverse event or a delay of the administration of the next dose due to toxicities for more than 14 days despite adequate medication or; drug-related grade 4 febrile neutropenia or; drug-related grade 4 anemia which cannot be adequately treated.
Phase 2: Overall Response Rate (ORR) | Up to 3.6 years
  ORR is defined as the sum of Complete remission (CR), CR with incomplete recovery (CRi), morphologic leukemia-free state (MLFS), partial remission (PR) at the ARGX-110 RP2D level that was established in Phase 1 according to established response criteria for Acute myeloid leukemia (AML).

SECONDARY OUTCOMES:
Phase 1 and Phase 2: Number of Participants with Adverse Events | Up to 3.6 years
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Phase 1 and Phase 2: Maximum Observed Concentration (Cmax) of ARGX-110 | Up to 3.6 years
  Cmax is the maximum observed concentration.
Phase 1 and Phase 2: Trough Concentration (Ctrough) of ARGX-110 | Up to 3.6 years
  Ctrough is defined as the observed serum concentration before dosing or at the end of the dosing interval.
Phase 1 and Phase 2: Area Under the Serum Concentration-Time Curve from Time Zero to Infinite (AUC[0-infinity]) of ARGX-110 | Up to 3.6 years
  AUC(0-infinity) is defined as area under the serum analyte concentration-time curve from time 0 to infinite time of ARGX-110.
Phase 1 and Phase 2: Area Under the Serum Concentration-Time Curve During the Dosing Interval (AUCtau) | Up to 3.6 years
  AUCtau is the area under the serum concentration-time curve during the dosing interval.
Phase 1 and Phase 2: Apparent Volume of Distribution (Vd/F) of ARGX-110 | Up to 3.6 years
  Vd/F is defined as Dose/[Lambda (z)*AUC (0-infinity)].
Phase 1 and Phase 2: Total Systemic Clearance (CL) of ARGX-110 | Up to 3.6 years
  CL is the total systemic clearance of drug after intravenous (IV) administration.
Phase 1 and Phase 2: Elimination Half-Life (t1/2) of ARGX-110 | Up to 3.6 years
  t1/2 is defined as the time measured for the serum concentration to decrease by 1 half of its original concentration.
Phase 1 and Phase 2: Number of Participants with Minimal Residual Disease (MRD) to ARGX-110 | Up to 3.6 years
  Minimal residual disease assessments will be performed on bone marrow aspirates and/or whole blood by flow cytometry.
Phase 1 and Phase 2: Number of Participants with Anti-drug Antibodies (ADA) to ARGX-110 | Up to 3.6 years
  Venous blood samples and bone marrow aspirate will be used to evaluate presence of anti-drug antibodies to ARGX-110. Participants with titer of confirmed positive samples for ARGX-110 antibodies will be reported.
Phase 1 and Phase 2: Number of Participants with Complete Remission (CR) | Up to 3.6 years
  Complete remission is defined as number of participants who have bone marrow blasts less than (<) 5 percent (%); absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count greater than (>) 1.0 * 10^9 per liter (L) (1000 per microliter [µL]); platelet count > 100 * 10^9/L (100.000/mc); independence of red cell transfusions.
Phase 1 and Phase 2: Number of Participants with CR with Incomplete Recovery (CRi) | Up to 3.6 years
  CRi is defined as number of participants who have all CR criteria except for residual neutropenia (< 1.0 * 10^9/L [1000/mc]) or thrombocytopenia (< 100 * 10^9/L [100.000/mc]).
Phase 1 and Phase 2: Number of Participants with Morphologic Leukemia-free State (MLFS) | Up to 3.6 years
  MLFS is defined as number of participants who have bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required.
Phase 1 and Phase 2: Number of Participants with Partial remission (PR) | Up to 3.6 years
  PR is defined as number of participants who have all hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
Phase 1 and Phase 2: Time to Response | Up to 3.6 years
  Time to response is defined as response measured from the time from first dose of study drug to date of response (CR, CRi, MLFS, PR).
Phase 1 and Phase 2: Duration of Response | Up to 3.6 years
  Duration of response is defined as the date of achievement of a response (CR, CRi, MLFS, PR) until the date of relapse.
Phase 1 and Phase 2: Relapse-Free Survival (RFS) | Up to 3.6 years
  RFS is defined as disease relapse or participant death from any cause; measured from the date of achievement of a remission (CR, CRi) until the date of relapse or death from any cause.
Phase 1 and Phase 2: Overall Survival (OS) | Up to 3.6 years
  OS is defined as death from any cause; measured from the date of first dose to the date of death from any cause.
Phase 1 and Phase 2: Number of Participants with 30 Day and 60 Day Mortality | 30 and/or 60 days after the first administration
  Number of participants with 30 Day and 60 Day Mortality will be reported.
Phase 1 and Phase 2: Number of Participants Achieving Transfusion Independence (TI) | Up to 3.6 years
  Number of participants reaching greater than or equal to (>=) 8 consecutive weeks without red blood cell (RBC-TI) and/or platelet (PLT-TI) transfusion. The first day of the >=8-week period with no transfusions is noted as the time at which participants first achieved TI.
Phase 1 and Phase 2: Time to Transfusion Independence | Up to 3.6 years
  Time until TI for RBC and/or PLT will be measured from the date of entry into a study to the first day of the 8-weeks period with no transfusions.
Phase 1 and Phase 2: Duration of Transfusion Independence | Up to 3.6 years
  Time between the last transfusion before the start of the TI period and the first transfusion after the start of the TI period, which occurred >=8 weeks later.
Phase 1 and Phase 2: Time to Neutrophil Recovery | Up to 3.6 years
  Time to neutrophil recovery will be calculated from number of days from Day 1 of commencing study treatment to first day neutrophils 0.5 * 10^9 per liter or 1.0 * 10^9 per liter.
Phase 1 and Phase 2: Time to Platelet Recovery | Up to 3.6 years
  Time to platelet recovery will be calculated from number of days from day 1 of commencing study treatment to first day neutrophils 50 * 10^9 per liter or 100 * 10^9 per liter.
Biomarker Assessment of ARGX-110 | Up to 3.6 years
  Biomarkers including CD70 and CD27 assessment will be performed on bone marrow aspirates and/or whole blood.
Phase 1: Levels of T, B and NK Cells | Up to 3.6 years
  Levels of T, B and NK cells will be reported by immunophenotyping (performed by flow cytometry or mass cytometry). .
Phase 1: Levels of B Cells | Up to 3.6 years
  Levels of B cells will be reported.
Phase 1: Levels of NK Cells | Up to 3.6 years
  Levels of NK cells will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- France (4):
  - Marseille
  - Paris
  - Pierre-Bénite
  - Toulouse
- Switzerland (3):
  - Aarau
  - Bern
  - Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Riether C, Pabst T, Hopner S, Bacher U, Hinterbrandner M, Banz Y, Muller R, Manz MG, Gharib WH, Francisco D, Bruggmann R, van Rompaey L, Moshir M, Delahaye T, Gandini D, Erzeel E, Hultberg A, Fung S, de Haard H, Leupin N, Ochsenbein AF. Targeting CD70 with cusatuzumab eliminates acute myeloid leukemia stem cells in patients treated with hypomethylating agents. Nat Med. 2020 Sep;26(9):1459-1467. doi: 10.1038/s41591-020-0910-8. Epub 2020 Jun 29. PMID 32601337